CLINICAL TRIAL: NCT02789774
Title: Randomised Controlled Trial on Surgical vs Non-surgical Treatment of Type II Odontoid Fracture Treatment in the Elderly
Brief Title: Uppsala Study on Odontoid Fracture Treatment in the Elderly
Acronym: USOFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USOFT
Record Dates: First submitted 2015-08-25; First posted 2016-06-03 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Spinal Fractures
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical treatment (Experimental): Stabilization of odontoid fracture with posterior fusion C1-C2
  Interventions: Procedure: Posterior fusion C1-C2
- Conservative treatment (Active Comparator): External stabilization of odontoid fracture with a rigid cervical collar for 3 months.
  Interventions: Procedure: Rigid cervical collar

INTERVENTIONS:
Procedure: Posterior fusion C1-C2 — Posterior access and screws in C1 (atlas) and C2 (axis) and fusion with addition of iliac crest bone graft. No postoperative collar.
  Other Names: Posterior atlantoaxial fusion
  Arms: Surgical treatment
Procedure: Rigid cervical collar — External immobilization of cervical spine in a rigid collar for 12 weeks.
  Other Names: cervical orthosis
  Arms: Conservative treatment

SUMMARY:
A multicenter randomized controlled trial is performed in Sweden (Uppsala, Malmo and Stockholm) comparing surgery with posterior C1-C2 fusion and conservative treatment with a rigid collar. Follow up will be performed up to one year after start of treatment registering EQ5D, NDI and cervical CT scans. Mortality will be documented during follow-up. All direct and indirect costs of treatment will be registered and used for cost-effectiveness analysis.

DETAILED DESCRIPTION:
50 patients, based on the following calculation of study size: The standard deviation for Neck Disability index, NDI, is just under 7, while "minimally clinical important difference" (MCID) is 7 points . That gives that 16 patients are needed in each group to get 80% power with a significance level of 5%. However, in the studied population the one year mortality rate is substantial, especially after a neck injury . In order to be able to draw conclusions from the study the investigators have elected to expand the study to 25 subjects in each group.

Follow up: 1w, 6w, 3m, 1y with CT, Questionaires: NDI, EQ5D. Bone density measurement at injury. Extension flexion x-ray after 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Acute displaced odontoid fracture type II according to Anderson and D'Alonzo, age 75 years or older. Displacement defined as 4 mm anterior translator displacement, any posterior translator displacement, or 10 degrees of angulation.

Exclusion Criteria:

* Any contraindication to surgery, anesthesia class ASA 4 or higher (Saklad 1941), severe senile dementia (defined as being admitted to a nursing home or hospital because of the dementia), anatomical or other prerequisites that makes an operation unsuitable.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2024-03 (Actual); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI questionnaire) | 1 year

SECONDARY OUTCOMES:
EQ5D questionnaire | 1 year
Number of participants that deceased after inclusion | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Lena Robinson, MD, Principal Investigator — Uppsala University Hospital
Locations (2):
- Sweden (2):
  - Uppsala University Hospital, Uppsala, Uppsala County
  - Malmö University Hospital, Malmo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kose et al. 2007
- [Background] Olerud et al. 1999
- [Derived] Robinson AL, Schmeiser G, Robinson Y, Olerud C. Surgical vs. non-surgical management of displaced type-2 odontoid fractures in patients aged 75 years and older: study protocol for a randomised controlled trial. Trials. 2018 Aug 22;19(1):452. doi: 10.1186/s13063-018-2690-8. PMID 30134944